CLINICAL TRIAL: NCT01459315
Title: Phase I, Open-Label Study in Healthy Male Subjects Describing GSK1349572 Exposure in Blood Plasma, Seminal Fluid and Rectal Mucosal Tissue Following Single and Multiple Dosing
Brief Title: GSK1349572 Exposure in Blood, Seminal Fluid, and Rectal Fluid and Tissue in Healthy Male Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: GlaxoSmithKline (Industry)
Responsible Party: Principal Investigator, Kristine Patterson, MD, Associate Professor, University of North Carolina, Chapel Hill
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 11-1733
Record Dates: First submitted 2011-10-21; First posted 2011-10-25 (Estimated); Last update posted 2013-07-04 (Estimated); Status verified 2013-07

CONDITIONS: Healthy
Keywords: Healthy; Male; GSK1349572; Dolutegravir; DTG; Integrase; HIV
MeSH Terms: interventions — dolutegravir

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- GSK1349572 (Experimental)
  Interventions: Drug: dolutegravir

INTERVENTIONS:
Drug: dolutegravir — Subjects will take a GSK1349572 (dolutegravir) 50mg tablet by mouth once daily for 8 days. GSK1349572 concentrations will be measured in blood plasma, seminal fluid, rectal fluid, and rectal tissue over 24 hours after a single dose and over two 24 hour periods once steady state is reached. Blood plasma will be collected pre-dose and 1, 2, 3, 4, 5, 6, 8, 12, 18, and 24 hours after dosing. Each subject will also provide a total of 9 seminal and rectal fluid samples and have 2 rectal tissue biopsies performed pre-dose or at 1, 3, 6, 12, 18, or 24 hours after receiving single or multiple doses.
  Other Names: GSK1349572; DTG

SUMMARY:
The purpose of this study is to describe drug concentrations in blood plasma, rectal fluid, rectal tissue, and seminal fluid in HIV negative men following single and multiple doses of an investigational HIV medication known as GSK1349572 (dolutegravir).

DETAILED DESCRIPTION:
The purpose of this study is to determine first dose and steady-state concentrations of GSK1349572 in seminal fluid, rectal mucosal fluid, and rectal tissue compared to blood plasma (BP) in HIV-1 negative males. GSK1349572 is an investigational next generation integrase inhibitor currently in Phase III trials. Understanding the concentrations of GSK1349572 in multiple male biological compartments will inform its role in preventing HIV infection by making an HIV-infected person less likely to transmit the virus, and protecting uninfected persons from acquiring the virus.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male subjects between the ages of 18 and 49 years, inclusive, with intact genital tract and gastrointestinal tract.
* Body Mass Index (BMI) of 18 to 30 kg/m2; and a total body weight greater than 50 kg (110 lbs).
* Evidence of a personally signed and dated informed consent document
* Willing and able to comply with all scheduled visits, treatment plan, laboratory tests, and other trial procedures.

Exclusion Criteria:

* Evidence or history of clinically significant hematological, renal, endocrine, pulmonary, gastrointestinal, cardiovascular, hepatic, psychiatric, neurologic, or allergic disease
* Subjects with a history of gastrectomy, colostomy, ileostomy, or any other procedure altering the gastrointestinal tract.
* Subjects with a history of vasectomy, prostatectomy, or any other procedure altering the male reproductive tract.
* Subjects with inflammatory bowel diseases (ulcerative colitis or Crohn's disease), irritable bowel syndrome, or other abnormalities of the colorectal mucosa, or significant colorectal symptom(s)
* Subject who is unwilling to refrain from any sexual activity for 72 hours before study visit Day 0 and until discharge from the study.
* Subject who is unwilling to refrain from rectal insertion of medical/recreation devices and products and from receptive anal intercourse, for 72 hours before study visit Day 0 and through 7 days after the last biopsy.
* History of febrile illness within 14 days prior to the first dose.
* Any condition possibly affecting drug absorption (eg, gastrectomy).
* A positive urine drug screen.
* A positive result for HIV, Hepatitis B surface antigen or Hepatitis B core antibody screening tests or anti-hepatitis C virus serology
* A positive test for syphilis, rectal gonorrhea, chlamydia, or HSV-2 (active lesions) at screening.
* Current alcohol consumption exceeding 14 drinks [1 drink = 5 ounces (150 mL) of wine or 12 ounces (360 mL) of beer or 1.5 ounces (45 mL) of spirits] per week or unwilling to abstain from alcohol use from 48 hours prior to the first dose of study medication until after the follow-up visit.
* History of regular use of tobacco- or nicotine-containing products exceeding an equivalent of 5 cigarettes per day within three months prior to screening or unwilling to abstain from cigarette smoking completely during visits.
* Treatment with an investigational drug within 4 months preceding the first dose of trial medication.
* Participated in a rectal biopsy study in the 12 months preceding the first dose of trial medication.
* Use of clinically significant prescription or non-prescription drugs within 7 days (or 14 days if the drug is a potential enzyme inducer) or 5 half-lives (whichever is longer) prior to the first dose of study medication
* Blood donation of approximately 1 pint (≥473 mL) within 56 days prior to dosing.
* History of sensitivity to heparin or heparin-induced thrombocytopenia.
* History of confirmed allergy to prescription or non-prescription products.
* Unable or unwilling to swallow oral medications.
* History of bleeding or clotting disorders including disseminated intravascular coagulation, hemophilia Henoch-Schönlein purpura (allergic purpura), hereditary hemorrhagic telangiectasia, thrombocytopenia, thrombophilia or Von Willebrand's disease.
* The subject's blood pressure is outside the range of 90-140/45-90 mmHg, or heart rate is outside the range of 45-100 bpm.
* Clinically significant abnormalities to pulse or conduction observed on ECG
* Unwilling or unable to comply with dietary restrictions
* Any other reason or condition that would make participation in the study unsafe, complicate interpretation of study outcome data, or interfere with achieving the study objectives.

Ages: 18 Years to 49 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 14 (Actual)
Dates: Start 2011-11; Primary Completion 2012-11 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Area under the concentration versus time curve (AUC) in blood plasma after a single dose | 24 hours
  The area under the concentration time curve will be determined from all sample collection time points over a 24 hour period. Sample collection for blood plasma will occur pre-dose, then 1, 2, 3, 4, 5, 6, 8, 12, 18, and 24 hours post-dose. AUCs will be determined for individual subjects and for all subjects combined following a single dose.
Peak concentration (Cmax) in blood plasma after a single dose | 24 hours
  Peak drug concentration in blood plasma after the first dose will be determined from samples taken pre-dose, then at 1, 2, 3, 4, 5, 6, 8, 12, 18, and 24 hours post-dose in each subject and across all subjects.
Area under the concentration versus time curve (AUC) in blood plasma at steady state | 24 hours
  The area under the concentration time curve will be determined from all sample collection time points over a 24 hour period. Sample collection for blood plasma will occur pre-dose, then 1, 2, 3, 4, 5, 6, 8, 12, 18, and 24 hours post-dose. AUCs will be determined for individual subjects and for all subjects combined at steady state.
Peak concentration (Cmax) in blood plasma at steady state | 24 hours
  Peak drug concentration in blood plasma at steady state will be determined from samples taken pre-dose, then at 1, 2, 3, 4, 5, 6, 8, 12, 18, and 24 hours post-dose in each subject and across all subjects.
Area under the concentration versus time curve (AUC) in seminal fluid after a single dose | 24 hours
  The area under the concentration time curve after a single dose will be determined from all sample collection time points over a 24 hour period for seminal fluid. Sample collection will occur pre-dose and at two time points per subject 1, 3, 6, 12, 18, or 24 hours post-dose. AUCs will be determined for all subjects combined.
Peak drug concentration (Cmax) in seminal fluid after a single dose | 24 hours
  Peak drug concentration in seminal fluid will be determined from samples taken pre-dose, then at 2 time points per subject 1, 3, 6, 12, 18, or 24 hours post-dose. Cmax will be determined for all subjects combined.
Area under the concentration versus time curve (AUC) for seminal fluid at steady state | 48 hours
  The area under the concentration time curve at steady state for seminal fluid will be determined from all sample collection time points over a 48 hour period for seminal fluid. Sample collection will occur at 1, 3, 6, 12, 18, or 24 hours post-dose over 48 hours with 3 collections per subject in each 24 hour period. AUCs will be determined for each subject and across all subjects.
Peak drug concentration (Cmax) for seminal fluid at steady state | 24 hours
  Peak drug concentration (Cmax) at steady state for seminal fluid will be determined from all sample collection time points over a 48 hour period. Sample collection will occur at 1, 3, 6, 12, 18, or 24 hours post-dose over 48 hours with 3 collections per subject in each 24 hour period. Cmax will be determined for each subject and across all subjects.
Area under the concentration versus time curve (AUC) for rectal fluid after a single dose | 24 hours
  The area under the concentration time curve after a single dose will be determined from all sample collection time points over a 24 hour period for rectal fluid. Sample collection will occur pre-dose and at two time points per subject 1, 3, 6, 12, 18, or 24 hours post-dose. AUCs will be determined for all subjects combined.
Peak drug concentration (Cmax) in rectal fluid after a single dose | 24 hours
  Peak drug concentration in rectal fluid will be determined from samples taken pre-dose, then at 2 time points per subject 1, 3, 6, 12, 18, or 24 hours post-dose. Cmax will be determined for all subjects combined.
Area under the concentration versus time curve (AUC) for rectal fluid at steady state | 48 hours
  The area under the concentration time curve at steady state for rectal fluid will be determined from all sample collection time points over a 48 hour period. Sample collection will occur at 1, 3, 6, 12, 18, or 24 hours post-dose over 48 hours with 3 collections per subject in each 24 hour period. AUCs will be determined for each subject and across all subjects.
Peak drug concentration (Cmax) for rectal fluid at steady state | 48 hours
  Peak drug concentration (Cmax) at steady state for rectal fluid will be determined from all sample collection time points over a 48 hour period. Sample collection will occur at 1, 3, 6, 12, 18, or 24 hours post-dose over 48 hours with 3 collections per subject in each 24 hour period. Cmax will be determined for each subject and across all subjects.
Area under the concentration versus time curve (AUC) for rectal tissue after a single dose | 24 hours
  The area under the concentration time curve for rectal tissue after a single dose will be determined from all sample collection time points over a 24 hour period. One sample collection will be performed per subject at either 1, 3, 6, 12, 18, or 24 hours post-dose and AUC will be determined for all subjects combined.
Peak drug concentration (Cmax) for rectal tissue after a single dose | 24 hours
  Peak drug concentration in rectal tissue after a single dose will be determined from all sample collection time points over a 24 hour period. One sample collection will be performed per subject at either 1, 3, 6, 12, 18, or 24 hours post-dose and Cmax will be determined for all subjects combined.
Area under the concentration versus time curve (AUC) for rectal tissue at steady state | 24 hours
  The area under the concentration time curve for rectal tissue at steady state will be determined from all sample collection time points over a 24 hour period. One sample collection will be performed per subject at either 1, 3, 6, 12, 18, or 24 hours post-dose and AUC will be determined for all subjects combined.
Peak drug concentration (Cmax) for rectal tissue at steady state | 24 hours
  Peak drug concentration in rectal tissue at steady state will be determined from all sample collection time points over a 24 hour period. One sample collection will be performed per subject at either 1, 3, 6, 12, 18, or 24 hours post-dose and Cmax will be determined for all subjects combined.
Area under the concentration versus time curve ratios after a single dose | 24 hours
  AUC ratios will be determined to compare blood plasma concentrations after a single dose with concentrations in rectal tissue, rectal fluid, and seminal fluid.
Area under the concentration time curve ratios at steady state | 24 hours
  AUC ratios will be determined to compare blood plasma concentrations at steady state with concentrations in rectal tissue, rectal fluid, and seminal fluid.
Accumulation ratio | 24
  Area under the concentration time curve (AUC) in each matrix at steady state will be compared to AUC after a single dose to determine accumulation ratios.

CONTACTS AND LOCATIONS:
Overall Officials: Kristine B Patterson, MD, Principal Investigator — University of North Carolina, Chapel Hill; Benjamin N Greener, PharmD, Study Director — University of North Carolina, Chapel Hill
Locations (1):
- University of North Carolina, Chapel Hill, Chapel Hill, North Carolina, United States